CLINICAL TRIAL: NCT05371483
Title: Cardiovascular and Cognitive Implications of Central Disorders of Hypersomnolence and Their Treatments
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Chad M. Ruoff, Principal Investigator, Mayo Clinic
Other Study IDs: 21-013321
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Narcolepsy; Idiopathic Hypersomnia
Keywords: Central Disorders of Hypersomnolence; Blood pressure; Cognitive function; narcolepsy; idiopathic hypersomnia
MeSH Terms: conditions — Narcolepsy; Idiopathic Hypersomnia | interventions — Blood Pressure Monitoring, Ambulatory; Actigraphy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Narcolepsy Type 1: Study participant will complete test(s) before and after taking a stable dose of a new/different hypersomnia medication. All hypersomnia medications will be prescribed and titrated by a clinical sleep specialist outside of this protocol.
  Interventions: Diagnostic Test: 24-hour Ambulatory Blood Pressure Monitoring; Diagnostic Test: Oculo-Cognitive Addition Test (OCAT)
- Narcolepsy Type 2: Study participant will complete test(s) before and after taking a stable dose of a new/different hypersomnia medication. All hypersomnia medications will be prescribed and titrated by a clinical sleep specialist outside of this protocol.
  Interventions: Diagnostic Test: 24-hour Ambulatory Blood Pressure Monitoring; Diagnostic Test: Oculo-Cognitive Addition Test (OCAT)
- Idiopathic Hypersomnia: Study participant will complete test(s) before and after taking a stable dose of a new/different hypersomnia medication. All hypersomnia medications will be prescribed and titrated by a clinical sleep specialist outside of this protocol.
  Interventions: Diagnostic Test: 24-hour Ambulatory Blood Pressure Monitoring; Diagnostic Test: Oculo-Cognitive Addition Test (OCAT)

INTERVENTIONS:
Diagnostic Test: 24-hour Ambulatory Blood Pressure Monitoring — Arm blood pressure cuff that will automatically inflate every 15-30 minutes to check blood pressure while awake and asleep over 24 hours. Patient will also complete a sleep diary and wear an actigraphy watch during this test.
  Other Names: Actigraphy; Sleep diary
Diagnostic Test: Oculo-Cognitive Addition Test (OCAT) — Tracks users' eye movements as they complete a simple mental addition test.

SUMMARY:
This is an observational study evaluating patients diagnosed with narcolepsy or idiopathic hypersomnia that have been prescribed a new/different hypersomnia treatment. The study is being done to better understand how hypersomnia treatment(s) impact blood pressure and cognitive function.

DETAILED DESCRIPTION:
This is an observational study evaluating how hypersomnia medications influence blood pressure and cognitive function in patients diagnosed with narcolepsy or idiopathic hypersomnia. Blood pressure will be assessed using 24-hour ambulatory blood pressure monitoring equipment. Cognitive function will be evaluated using the Oculo-Cognitive Addition Test (OCAT). Both tests will performed at baseline (e.g., before starting a new hypersomnia medication) and after taking a stable dose of the new hypersomnia medication for at least three months. All medications will be prescribed by a clinical sleep specialist as part of routine medical care and covered by subject's health insurance plan (i.e., no medications are dispensed/titrated/paid for by the study investigators/trial).

The 24-hour ambulatory blood pressure test will be setup in person by staff. During the blood pressure test, the study participant will also complete a sleep diary and wear an actigraphy watch to track activity and sleep-wake cycle. The 24-hour ambulatory blood pressure test will be programmed to inflate a blood pressure cuff placed around the arm every 15 - 30 minutes.

The OCAT test, which takes approximately 15-20 minutes to complete, will be completed in person as well.

Each study participant may complete one or both tests. Each study participant may complete more than two assessments (e.g., patient that has been prescribed a second hypersomnia medication). If a patient presents already taking a medication of interest at baseline for at least the last 3 months then the participant may undergo baseline assessment(s) while taking respective medication(s).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with narcolepsy or idiopathic hypersomnia according to International Classification of Sleep Disorders, third edition
* Age 18 - 75 years
* BMI between 18 and 40 kg/m2
* Prescribed a medication of interest (e.g., sodium oxybate, low sodium oxybate, pitolisant, modafinil/armodafinil, solriamfetol, traditional stimulant(s)) by a clinical sleep specialist as part of routine medical care.
* Subject must be willing to postpone starting medication until after completion of baseline assessment(s).
* If subject has been taking a prescribed hypersomnia medication(s) at a stable dose for at least 3 months and has been prescribed a new medication, then subject may complete baseline assessment(s) while taking initial hypersomnia medication(s) before starting new medication.

Exclusion Criteria:

* Any change to medication(s) within the last 45 days
* History of chronic alcohol or drug abuse within the prior 12 months
* Heart failure, history of severe hypertension, or other cardiovascular disease compromising the patient's wellbeing or ability to participate in this study
* Use of any sleep apnea treatment (e.g., Positive Airway Pressure (PAP) therapy, oral appliance therapy, etc.) within 45 days of baseline assessment visit
* Participation in another study of an investigational drug within the 28 days prior to screening visit or currently
* Pregnancy and/or breast-feeding
* Subjects who, in the opinion of the Investigator, may not be suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with narcolepsy or idiopathic hypersomnia that have been prescribed but not yet started a new/different hypersomnia medication.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in mean 24-hour ambulatory blood pressure | Baseline, at least 3 months
  Change in 24-hour ambulatory blood pressure from baseline (pre-treatment) to after taking a stable dose of medication for at least 3 months

SECONDARY OUTCOMES:
Change in Oculo-Cognitive Addition Test (OCAT) completion time | Baseline, at least 3 months
  Change in OCAT completion time from baseline (pre-treatment) to after taking a stable dose of medication for at least 3 months (post-treatment)
Change in mean daytime and nighttime 24-hour ambulatory blood pressure | Baseline, at least 3 months
  Change in mean daytime and nighttime 24-hour ambulatory blood pressure from baseline (pre-treatment) to after taking a stable dose of medication for at least 3 months (post-treatment)
Change in 24-hour ambulatory blood pressure diurnal pattern (dipper versus non-dipper) | Baseline, at least 3 months
  Change in 24-hour ambulatory blood pressure diurnal pattern (dipper versus non-dipper) from baseline (pre-treatment) to after taking a stable dose of medication for at least 3 months (post-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Ruoff, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No